CLINICAL TRIAL: NCT02855931
Title: A Randomized Controlled Trial Comparing Partial Resection Versus Preservation of the Middle Turbinate in Surgery for Chronic Rhinosinusitis With Polyposis (CRSwP)
Brief Title: Study to Compare Resection Versus Preservation of the Middle Turbinate in Surgery for Nasal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie Bussières, Otolaryngologist - head and neck surgeon, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-1318
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Nasal Polyps; Sinusitis
MeSH Terms: conditions — Nasal Polyps; Sinusitis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Middle turbinate resection (Experimental): Resection of one middle turbinate
  Interventions: Procedure: Middle turbinate resection
- Middle turbinate preservation (No Intervention): Preservation of one middle turbinate

INTERVENTIONS:
Procedure: Middle turbinate resection
  Arms: Middle turbinate resection

SUMMARY:
Endoscopic sinus surgery (ESS) has become the standard of care for patients suffering of chronic rhinosinusitis with nasal polyposis (CRSwP) who have failed medical therapy. The goal of surgery is now to widely marsupialize the sinus cavities in order to optimize topical steroid irrigation treatment in the postoperative period. With that being said, the true extent of surgery needed for optimal patient outcome has yet to be elucidated. More specifically, in the last 30 years, people have argued about the best way to manage the middle turbinate. Some state that it should be preserved at all times to protect the sinus cavities from inhaled irritants and allergens and keep this surgical landmark untouched for future surgeries. On the other hand, there are defenders of routine resection of this turbinate, whether it is affected by polypoid changes or not. Many studies have looked at the potential risks of resecting the middle turbinates such as iatrogenic frontal sinusitis, anosmia, or atrophic rhinitis but the more recent literature does not show such significant associations. A recent topic of debate is whether partial removal of the anterior and inferior portion of the middle turbinate affects nasal polyps recurrence or improves long-term outcomes by further facilitation of post-operative topical therapies. Some retrospective data has shown that its resection could prolong the time before the need for revision surgery and improve both endoscopic and olfaction scores. A few prospective studies have also been published but unfortunately none of these were randomized, thus introducing a significant selection bias. Thus, there is a need for a formal randomized, controlled trial to elucidate this question.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis with nasal polyposis
* Obtained consent for bilateral complete endoscopic sinus surgery (maxillary antrostomy, complete sphenoethmoidectomy and frontal recess surgery)
* Primary or revision surgery

Exclusion Criteria:

* Allergic fungal sinusitis
* Patients with previous surgery which included partial or complete middle turbinectomy, uni- or bilateral
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the PeriOperative Sinus Endoscopy (POSE) score | Postoperative evaluations at 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bussières, MD, FRCSC, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Département de chirurgie, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Hudon MA, Wright ED, Fortin-Pellerin E, Bussieres M. Resection versus preservation of the middle turbinate in surgery for chronic rhinosinusitis with nasal polyposis: a randomized controlled trial. J Otolaryngol Head Neck Surg. 2018 Nov 8;47(1):67. doi: 10.1186/s40463-018-0313-8. PMID 30409178